CLINICAL TRIAL: NCT04320888
Title: NCI-COG Pediatric MATCH (Molecular Analysis for Therapy Choice) - Phase 2 Subprotocol of LOXO-292 in Patients With Tumors Harboring RET Gene Alterations
Brief Title: Selpercatinib for the Treatment of Advanced Solid Tumors, Lymphomas, or Histiocytic Disorders With Activating RET Gene Alterations, a Pediatric MATCH Treatment Trial
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Children's Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2020-01756; NCI-2020-01756 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); APEC1621N (Other: Children's Oncology Group); APEC1621N (Other: CTEP); U10CA180886 (NIH)
Record Dates: First submitted 2020-03-24; First posted 2020-03-25 (Actual); Results first posted 2025-11-06 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-10

CONDITIONS: Hematopoietic and Lymphatic System Neoplasm; Recurrent Ependymoma; Recurrent Ewing Sarcoma; Recurrent Hepatoblastoma; Recurrent Histiocytic and Dendritic Cell Neoplasm; Recurrent Langerhans Cell Histiocytosis; Recurrent Lymphoma; Recurrent Malignant Germ Cell Tumor; Recurrent Malignant Glioma; Recurrent Malignant Solid Neoplasm; Recurrent Medulloblastoma; Recurrent Neuroblastoma; Recurrent Non-Hodgkin Lymphoma; Recurrent Osteosarcoma; Recurrent Peripheral Primitive Neuroectodermal Tumor; Recurrent Rhabdoid Tumor; Recurrent Rhabdomyosarcoma; Recurrent Soft Tissue Sarcoma; Recurrent WHO Grade 2 Glioma; Refractory Ependymoma; Refractory Ewing Sarcoma; Refractory Hepatoblastoma; Refractory Histiocytic and Dendritic Cell Neoplasm; Refractory Langerhans Cell Histiocytosis; Refractory Lymphoma; Refractory Malignant Germ Cell Tumor; Refractory Malignant Glioma; Refractory Malignant Solid Neoplasm; Refractory Medulloblastoma; Refractory Neuroblastoma; Refractory Non-Hodgkin Lymphoma; Refractory Osteosarcoma; Refractory Peripheral Primitive Neuroectodermal Tumor; Refractory Rhabdoid Tumor; Refractory Rhabdomyosarcoma; Refractory Soft Tissue Sarcoma; Refractory WHO Grade 2 Glioma; Wilms Tumor
MeSH Terms: conditions — Ependymoma; Sarcoma, Ewing; Hepatoblastoma; Histiocytosis, Langerhans-Cell; Lymphoma; Glioma; Medulloblastoma; Neuroblastoma; Lymphoma, Non-Hodgkin; Osteosarcoma; Neuroectodermal Tumors, Primitive, Peripheral; Rhabdoid Tumor; Rhabdomyosarcoma; Sarcoma; Wilms Tumor | interventions — Magnetic Resonance Spectroscopy; Nuclear Medicine Department, Hospital; selpercatinib; X-Rays; Phantoms, Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (selpercatinib) (Experimental): Patients receive selpercatinib PO BID on days 1-28. Treatment repeats every 28 days for up to 26 cycles (2 years) in the absence of disease progression or unacceptable toxicity. Patients may also undergo PET, CT, MRI, PET/CT, PET/MRI, and/or CT/MRI, scintigraphy, and x-ray imaging throughout the trial.
  Interventions: Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Procedure: Radionuclide Imaging; Drug: Selpercatinib; Procedure: X-Ray Imaging

INTERVENTIONS:
Procedure: Computed Tomography — Undergo CT, PET/CT, and/or CT/MRI
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI, PET/MRI, and/or CT/MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Positron Emission Tomography — Undergo PET, PET/CT, and/or PET/MRI
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Procedure: Radionuclide Imaging — Undergo scintigraphy
  Other Names: NM; Nuclear Medicine; nuclear medicine scan; radioimaging; Radionuclide Scanning; Scan; Scintigraphy
Drug: Selpercatinib — Given PO
  Other Names: LOXO 292; LOXO-292; LOXO292; RET Kinase Inhibitor LOXO-292; Retevmo; Retsevmo; WHO 10967
Procedure: X-Ray Imaging — Undergo x-ray imaging
  Other Names: Conventional X-Ray; Diagnostic Radiology; Medical Imaging, X-Ray; Plain film radiographs; Radiographic Imaging; Radiographic imaging procedure (procedure); Radiography; RG; Static X-Ray; X-Ray

SUMMARY:
This phase II pediatric MATCH treatment trial studies how well selpercatinib works in treating patients with solid tumors that may have spread from where they first started to nearby tissue, lymph nodes, or distant parts of the body (advanced), lymphomas, or histiocytic disorders that have activating RET gene alterations. Selpercatinib may block the growth of cancer cells that have specific genetic changes in an important signaling pathway (called the RET pathway) and may reduce tumor size.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the objective response rate (ORR; complete response + partial response) in pediatric patients treated with selpercatinib (LOXO-292) with advanced solid tumors (including central nervous system [CNS] tumors), lymphomas or histiocytic disorders that harbor activating genetic alterations in the RET pathway.

SECONDARY OBJECTIVES:

I. To estimate the progression free survival in pediatric patients treated with selpercatinib (LOXO-292) with advanced solid tumors (including CNS tumors), lymphomas or histiocytic disorders that harbor activating genetic alterations in the RET pathway.

II. To obtain information about the tolerability of selpercatinib (LOXO-292) in children and adolescents with relapsed or refractory cancer.

EXPLORATORY OBJECTIVE:

I. To explore approaches to profiling changes in tumor genomics over time through evaluation of circulating tumor deoxyribonucleic acid (DNA).

OUTLINE:

Patients receive selpercatinib orally (PO) twice daily (BID) on days 1-28 on study. Treatment repeats every 28 days for up to 26 cycles (2 years) in the absence of disease progression or unacceptable toxicity. Patients may also undergo positron emission tomography (PET), computed tomography (CT), magnetic resonance imaging (MRI), PET/CT, PET/MRI, and/or CT/MRI, scintigraphy, and x-ray imaging throughout the trial.

After completion of study treatment, patients are followed for 30 days, then periodically thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have enrolled onto APEC1621SC and must have been given a treatment assignment to MATCH to APEC1621N based on the presence of an actionable mutation
* Patients must be >= 12 months and =< 21 years of age at the time of study enrollment
* Patients must have radiographically measurable disease at the time of study enrollment. Patients with neuroblastoma who do not have measurable disease but have metaiodobenzylguanidine (MIBG) positive (+) evaluable disease are eligible. Measurable disease in patients with CNS involvement is defined as any lesion that is at minimum 10 mm in one dimension on standard MRI or CT

  * Note: The following do not qualify as measurable disease:

    * Malignant fluid collections (e.g., ascites, pleural effusions)
    * Bone marrow infiltration except that detected by MIBG scan for neuroblastoma
    * Lesions only detected by nuclear medicine studies (e.g., bone, gallium or positron emission tomography [PET] scans) except as noted for neuroblastoma
    * Elevated tumor markers in plasma or cerebral spinal fluid (CSF)
    * Previously radiated lesions that have not demonstrated clear progression post radiation
    * Leptomeningeal lesions that do not meet the measurement requirements for Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
* Karnofsky >= 50% for patients > 16 years of age and Lansky >= 50 for patients =< 16 years of age. Note: Neurologic deficits in patients with CNS tumors must have been relatively stable for at least 7 days prior to study enrollment. Patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score
* Patients must have fully recovered from the acute toxic effects of all prior anti-cancer therapy and must meet the following minimum duration from prior anti-cancer directed therapy prior to enrollment. If after the required timeframe, the numerical eligibility criteria are met, e.g. blood count criteria, the patient is considered to have recovered adequately

  * Cytotoxic chemotherapy or other anti-cancer agents known to be myelosuppressive.

    * >= 21 days after the last dose of cytotoxic or myelosuppressive chemotherapy (42 days if prior nitrosourea)
  * Anti-cancer agents not known to be myelosuppressive (e.g. not associated with reduced platelet or absolute neutrophil [ANC] counts): >= 7 days after the last dose of agent.
  * Antibodies: >= 21 days must have elapsed from infusion of last dose of antibody, and toxicity related to prior antibody therapy must be recovered to grade =< 1
  * Corticosteroids: If used to modify immune adverse events related to prior therapy, >= 14 days must have elapsed since last dose of corticosteroid
  * Hematopoietic growth factors: >= 14 days after the last dose of a long-acting growth factor (e.g. pegfilgrastim) or 7 days for short-acting growth factor. For growth factors that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur. The duration of this interval must be discussed with the study chair and the study-assigned research coordinator
  * Interleukins, interferons and cytokines (other than hematopoietic growth factors): >= 21 days after the completion of interleukins, interferon or cytokines (other than hematopoietic growth factors)
  * Stem cell infusions (with or without total body irradiation [TBI]):

    * Allogeneic (non-autologous) bone marrow or stem cell transplant, or any stem cell infusion including donor lymphocyte infusion (DLI) or boost infusion: >= 84 days after infusion and no evidence of graft versus host disease (GVHD)
    * Autologous stem cell infusion including boost infusion: >= 42 days
  * Cellular therapy: >= 42 days after the completion of any type of cellular therapy (e.g. modified T cells, natural killer [NK] cells, dendritic cells, etc.)
  * Radiation therapy (XRT)/external beam irradiation including protons: >= 14 days after local XRT; >= 150 days after TBI, craniospinal XRT or if radiation to >= 50% of the pelvis; >= 42 days if other substantial bone marrow (BM) radiation

    * Note: Radiation may not be delivered to "measurable disease" tumor site(s) being used to follow response to subprotocol treatment
  * Radiopharmaceutical therapy (e.g., radiolabeled antibody, 131I-MIBG): >= 42 days after systemically administered radiopharmaceutical therapy
  * Patients must not have received prior exposure to selpercatinib (LOXO-292) or other specific RET inhibitors
* For patients with solid tumors without known bone marrow involvement (within 7 days prior to enrollment):

  * Peripheral absolute neutrophil count (ANC) >= 1000/mm^3
* For patients with solid tumors without known bone marrow involvement (within 7 days prior to enrollment):

  * Platelet count >= 100,000/mm^3 (transfusion independent, defined as not receiving platelet transfusions for at least 7 days prior to enrollment)
* Patients with known bone marrow metastatic disease will be eligible for study provided they meet the blood counts (may receive transfusions provided they are not known to be refractory to red cell or platelet transfusions). These patients will not be evaluable for hematologic toxicity
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70 ml/min/1.73 m^2 (within 7 days prior to enrollment) or a serum creatinine based on age/gender as follows (within 7 days prior to enrollment):

  * Age: Maximum serum creatinine (mg/dL)

    * 1 to < 2 years: male (0.6), female (0.6)
    * 2 to < 6 years: male (0.8), female (0.8)
    * 6 to < 10 years: male (1), female (1)
    * 10 to < 13 years: male (1.2), female (1.2)
    * 13 to < 16 years: male (1.5), female (1.4)
    * >= 16 years: male (1.7), female (1.4)
* Bilirubin (sum of conjugated + unconjugated) =< 1.5 x upper limit of normal (ULN) for age (within 7 days prior to enrollment)
* Serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) =< 135 U/L. (within 7 days prior to enrollment) (For the purpose of this study, the ULN for SGPT is 45 U/L.)
* Serum albumin >= 2 g/dL (within 7 days prior to enrollment)
* Corrected QT (QTc) interval =< 480 milliseconds (within 7 days prior to enrollment)
* All patients and/or their parents or legally authorized representatives must sign a written informed consent. Assent, when appropriate, will be obtained according to institutional guidelines

Exclusion Criteria:

* Pregnant or breast-feeding women will not be entered on this study due to risks of fetal and teratogenic adverse events as seen in animal/human studies. Pregnancy tests must be obtained in girls who are post-menarchal. Males or females of reproductive potential may not participate unless they have agreed to use two (2) highly effective contraceptive method for the duration of study treatment and for at least 2 weeks after the last dose of selpercatinib (LOXO-292). Male study participants are to refrain from sperm donation during treatment and for 2 weeks after the last dose of selpercatinib (LOXO-292)
* Patients receiving corticosteroids who have not been on a stable or decreasing dose of corticosteroid for at least 7 days prior to enrollment are not eligible. If used to modify immune adverse events related to prior therapy, >= 14 days must have elapsed since last dose of corticosteroid
* Patients who are currently receiving another investigational drug are not eligible
* Patients who are currently receiving other anti-cancer agents are not eligible
* Patients who are receiving cyclosporine, tacrolimus or other agents to prevent graft-versus-host disease post bone marrow transplant are not eligible for this trial
* Patients who are currently receiving drugs that are moderate or strong inducers or inhibitors of CYP3A4 are not eligible. Strong inducers or inhibitors of CYP3A4 should be avoided from 14 days prior to enrollment to the end of the study. Note: CYP3A4 inducing anti-epileptic drugs and dexamethasone for CNS tumors or metastases, on a stable dose, are allowed
* Proton pump inhibitors (PPIs), H2 receptor antagonists and antacids: Concomitant use of PPIs during selpercatinib (LOXO-292) therapy should be avoided if feasible. If co-administration of selpercatinib and PPI is necessary, administer selpercatinib with a meal. If H2 receptor antagonist is necessary, administer selpercatinib 2 hours before or 10 hours after H2 receptor antagonist administration. If antacid use is necessary, administer selpercatinib 2 or more hours before or 2 or more hours after antacid administration
* Patients who have major surgery within 14 days prior to cycle 1 day 1 (C1D1) are not eligible. (Central line placement or subcutaneous port placement is not considered major surgery)
* Patients with known clinically significant active malabsorption syndrome or other condition likely to affect gastrointestinal absorption of selpercatinib (LOXO-292) are excluded
* Patients with known hypersensitivity to any of the components of the investigational agent, LOXO 292 are excluded
* Patients with uncontrolled hypertension are excluded
* Patients with uncontrolled symptomatic hyperthyroidism and hypothyroidism (i.e. the patient required a modification to current thyroid medication in 7 days prior to enrollment) are excluded
* Patients with uncontrolled symptomatic hypercalcemia and hypocalcemia are excluded
* Patients who have an uncontrolled infection are not eligible
* Patients who have received a prior solid organ transplantation are not eligible
* Patients who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study are not eligible

Ages: 12 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2021-05-03 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2026-06-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea T Franson, Principal Investigator — Children's Oncology Group
Locations (174):
- United States (172):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Banner Children's at Desert, Mesa, Arizona
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Kaiser Permanente Downey Medical Center, Downey, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Mattel Children's Hospital UCLA, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - Naval Medical Center -San Diego, San Diego, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center, Torrance, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - Miami Cancer Institute, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Tampa General Hospital, Tampa, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Saint Mary's Medical Center, West Palm Beach, Florida
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Ascension Saint Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Maine Children's Cancer Program, Scarborough, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Michigan State University, East Lansing, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Corewell Health Children's, Royal Oak, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Albany Medical Center, Albany, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Mission Hospital, Asheville, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Saint Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - T C Thompson Children's Hospital, Chattanooga, Tennessee
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - The Children's Hospital at TriStar Centennial, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - El Paso Children's Hospital, El Paso, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - UMC Cancer Center / UMC Health System, Lubbock, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Naval Medical Center - Portsmouth, Portsmouth, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - West Virginia University Healthcare, Morgantown, West Virginia
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Perth Children's Hospital, Perth, Western Australia, Australia
- University Pediatric Hospital, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Selpercatinib)
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Data not provided as confidentiality is an issue.
Arm/Group | Treatment (Selpercatinib)
Number analyzed (Participants) | 0
Age, Categorical
Age, Continuous [unit: years]
Sex: Female, Male
Ethnicity (NIH/OMB)
Race (NIH/OMB)

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (Complete Response + Partial Response) in Pediatric Patients Treated With Selpercatinib (LOXO-292)
Description: A responder is defined as a patient who achieves a best response of partial response or complete response on the study. Response rates will be calculated as the percent of evaluable patients who are responders. The revised Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1) was used to determine response and progression in this study, with specific criteria outlined for the different subtypes of tumors (e.g., 2-dimensional measurements for central nervous system [CNS] tumors).
Time Frame: Up to 2 years from study entry
Measure: Number; unit: percentage of participants
Arm/Group | Treatment (Selpercatinib)
Number analyzed (Participants) | 1
percentage of participants | 100

2. Secondary Outcome: Progression-free Survival (PFS)
Description: The Kaplan-Meier method will be used to estimate the 6 month PFS. PFS is defined as time from initiation of protocol treatment to disease progression, recurrence, death from any cause, or date of last contact.
Time Frame: Up to 6 months from study entry
Measure: Number; unit: percentage of participants
Arm/Group | Treatment (Selpercatinib)
Number analyzed (Participants) | 1
percentage of participants | 100

3. Secondary Outcome: Percentage of Patients Experiencing Grade 3 or 4 Adverse Events
Description: Evaluated by Common Terminology Criteria for Adverse Events version 5. Any eligible patient who receives at least one dose of protocol therapy will be considered in the evaluation of toxicity.
Time Frame: Up to 2 years from study entry
Measure: Number; unit: percentage of participants
Arm/Group | Treatment (Selpercatinib)
Number analyzed (Participants) | 1
percentage of participants | 0

4. Other Pre Specified Outcome: Profiling Changes in Tumor Genomics
Description: Will explore approaches to the profiling changes in tumor genomics over time through evaluation of circulating tumor deoxyribonucleic acid. A descriptive analysis will be performed and will be summarized with simple summary statistics. All of these analyses will be descriptive in nature.
Time Frame: Up to time of disease progression or end of protocol therapy
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 2 years from study entry
Description: Adverse event reporting is collected routinely using case report forms. The SAE table reflects NCI Common Terminology Criteria for Adverse Events (CTCAEs) submitted by the institution via expedited reporting (NCI AdEERs / CAeRs). All remaining CTCAEs collected by means other than expedited reporting are non-serious and are reported in the "AE Other" table. All-Cause Mortality includes all deaths collected on the study. Ineligible patients are excluded from reporting of adverse events.
Arm/Group | Treatment (Selpercatinib)
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Selpercatinib) (N=1)
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Dry mouth (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Stomach pain (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 1
Infections and infestations - Other, specify (Infections and infestations) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1

LIMITATIONS AND CAVEATS:
This study had significant limitations as it did not reach the target number of participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-10-28): https://cdn.clinicaltrials.gov/large-docs/88/NCT04320888/Prot_SAP_000.pdf
  • Informed Consent Form (2022-10-28): https://cdn.clinicaltrials.gov/large-docs/88/NCT04320888/ICF_001.pdf